CLINICAL TRIAL: NCT06950255
Title: Effect of a 3-week Program of Cane Training and Use on Gait of Individuals With Parkinson's Disease: Protocol for a Randomized Controlled Trial
Brief Title: Effect of Training and Use of Cane on Gait in Individuals With Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Pró-reitoria de Pesquisa da Universidade Federal de Minas Gerais (Unknown)
Responsible Party: Principal Investigator, Christina Danielli Coelho de Morais Faria, Principal Investigator, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE: 75158123.2.0000.5149
Record Dates: First submitted 2025-04-22; First posted 2025-04-30 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease
Keywords: assistive device; canes; mobility; gait
MeSH Terms: conditions — Parkinson Disease | interventions — Canes; Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The collection will be performed by a previously trained examiner, blinded to the allocation of groups. All participants will be instructed not to comment on information about the training received. The therapist responsible for delivering the intervention will be blinded to the results of participants' assessments All statistical analyzes will be performed by an independent examiner, blinded to all procedures performed in the study, including with regard to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): After allocation, individuals in the experimental group will receive cane usage training, provided in four sessions lasting 40 minutes each, spaced over a period of 15 to 22 days. Additionally, they will be instructed and encouraged to use the cane in their daily mobility activities, both indoors and outdoors, starting from the first day of training. To monitor adherence, individuals will receive a diary to record on which occasions and for how long they used the cane during mobility activities. To enhance adherence, participants will receive telephone follow-ups between sessions aimed at monitoring and encouraging device use.
  Interventions: Device: Cane
- Time and attention control group (Sham Comparator): To ensure a comparable amount of attention received, individuals in the control group will receive an intervention involving global stretching of the upper and lower limbs and health education. The intervention will be provided in four sessions lasting 40 minutes each, spaced for 15 to 22 days. Additionally, individuals allocated to the control group will be instructed not to start using any assistive device during the study period and encouraged to perform stretching daily at home from the first day of training. To monitor adherence, individuals will receive a diary to record stretching exercises performed daily. To enhance adherence, participants will receive telephone follow-ups between sessions aimed at monitoring and encouraging the performance of the stretching exercises.
  Interventions: Other: static stretching and health education

INTERVENTIONS:
Device: Cane — Individuals will receive a single-point cane, individually adjusted to maintain each individual's elbow at approximately 30 degrees of flexion. Participants will be instructed to use the device on dominant side or the side with less impairment. The training with the cane will be carried out by a trained physiotherapist. The training protocol will include gait training with the cane on different surfaces and speeds. At the beginning of each training session, individuals will have the opportunity to address any questions they may have about using a cane in their daily life context.
  Individuals will be re-evaluated after the end of the training sessions. After revaluation, the canes will be left with participants who will be instructed as follows: "Feel free to use the cane at any time as needed." Another diary will be provided for the participant to record the use of the device after the end of the intervention
  Arms: Experimental group
Other: static stretching and health education — The intervention for the control group will consist of 20 minutes of global static stretching and 20 minutes of guidance on general health care. The stretches will be performed in three sets of 30 seconds each, targeting different muscle groups. If a participant is unable to perform the self-stretches, the researchers responsible for implementing the intervention will provide assistance. The health education component will cover information on Parkinson's disease (PD) and fall prevention.
  The intervention will be offered by the same physiotherapist responsible for training the experimental group. Individuals will be re-evaluated after the end of the training sessions. After revaluation, the participants will be instructed as follows: "Feel free to continue stretching exercises and use the health information discussed as needed." Another diary will be provided for the participant to record the stretching exercises performed after the end of the intervention.
  Arms: Time and attention control group

SUMMARY:
Introduction: Although individuals with Parkinson's disease (PD) commonly use assistive devices, the effects of these devices on gait remain poorly understood. Furthermore, previous studies on this topic only investigated the immediate effects of device usage, and the investigated outcomes were predominately performance-based neglecting participant-centered outcomes.

Objective: To investigate the effect of cane training and use on gait speed (primary outcome), gait confidence, cadence, step length, functional mobility, freezing of gait, fear of falls and satisfaction with the use of a cane (secondary outcomes) in individuals with PD.

Methods: A double-blind, randomized controlled trial with intention-to-treat and per-protocol analysis will be carried out. A total of 26 individuals with PD will be recruited based on the following inclusion criteria: age ≥ 40 years, diagnosis of idiopathic PD, classification between stages II to IV on the modified Hoehn & Yahr Scale, stable use of anti-parkinsonian pharmacological therapy, ability to walk independently with a walking speed ≤ 1.1 m/s (defined to screen individuals with gait impairments), and ability to use a single-point cane during walking without regular use of any type of assistive device since the diagnosis of PD. Participant will be randomly divided into two groups that will receive: (1) cane training and use (experimental group) or (2) global stretches and health education (time and attention-controlled group). The intervention will be provided in four sessions lasting 40 minutes each, spaced over 15 to 22 days. Additionally, individuals will be instructed to use a cane (experimental group) or perform stretching exercises (time and attention-controlled group) daily, starting from the first day of training. Assessments will be conducted at the beginning of the study (week 0), post-intervention (after the 3-week intervention), and one month after the cessation of the intervention (8-week follow-up). The primary outcomes is gait speed. Secondary outcomes include gait confidence, cadence, step length, functional mobility, freezing of gait, fear of falls, and satisfaction with the use of a cane. Between-group differences will be measured using a two-way repeated measures ANOVA, considering baseline, post-intervention, and follow-up assessments, following both intention-to-treat and per-protocol approaches (α=0.05).

Conclusions: The results of the present study will provide information about the effects of cane training and use on the gait of individuals with PD who will have the opportunity to use the cane in their real-life context.

DETAILED DESCRIPTION:
A non-probabilistic sample will be recruited from the community. Individuals will be included according to the following criteria: age ≥ 40 years; diagnosis of idiopathic PD confirmed by a neurologist; classification between stages II to IV of the modified Hoehn & Yahr Scale (HY); use of anti-parkinsonian medication with stable pharmacological therapy for at least 6 months; ability to walk independently in a 14-meter corridor with a walking speed ≤ 1.1 m/s (defined to screen individuals with gait impairments); ability to use a single-point cane during walking correctly and safely without regular use of any type of assistive device since the diagnosis of PD. Individuals with cognitive impairment, using deep brain stimulation, or who present any other condition that may compromise the test performance will be excluded. Two individuals with PD were involved as collaborators in this study to contribute to the relevance of the research through the inclusion of patient perspectives.

After baseline assessments individuals will be randomly allocated into the experimental and control groups. After allocation, all individuals will be instructed to maintain their usual healthcare routines.

Individuals in the experimental group will receive cane usage training, provided in four sessions lasting 40 minutes each, spaced over a period of 15 to 22 days. Additionally, they will be instructed and encouraged to use the cane in their daily mobility activities, both indoors and outdoors, starting from the first day of training. To monitor adherence, individuals will receive a diary to record on which occasions and for how long they used the cane during gait activities. To enhance adherence, participants will receive telephone follow-ups between sessions aimed at monitoring and encouraging device use. Individuals will be re-evaluated after the end of the training sessions. After revaluation, the canes will be left with participants who will be instructed as follows: "Feel free to use the cane at any time as needed." Another diary will be provided for the participant to record the use of the device after the end of the intervention.

To ensure a comparable amount of attention received, individuals in the control group will receive an intervention involving global stretching of the upper and lower limbs and health education. The intervention will be provided in four sessions lasting 40 minutes each, spaced for 15 to 22 days. Additionally, individuals allocated to the control group will be instructed not to start using any assistive device during the study period and encouraged to perform stretching daily at home from the first day of training. To monitor adherence, individuals will receive a diary to record stretching exercises performed daily. To enhance adherence, participants will receive telephone follow-ups between sessions aimed at monitoring and encouraging the performance of the stretching exercises.The intervention will be offered by the same physiotherapist responsible for training the experimental group. Individuals will be re-evaluated after the end of the training sessions. After revaluation, the participants will be instructed as follows: "Feel free to continue stretching exercises and use the health information discussed as needed." Another diary will be provided for the participant to record the stretching exercises performed after the end of the intervention.

The primary outcomes is gait speed. Secondary outcomes include gait confidence, cadence, step length, functional mobility, freezing of gait , fear of falls, and satisfaction with the use of a cane. Adverse events will be monitored throughout the intervention. They are defined as any unexpected medical issue related to the intervention-such as pain, falls, or exercise intolerance-that requires hospitalization or additional treatment.

The sample size was calculated based on a clinically meaningful difference of 0.22 m/s and a standard deviation of 0.15 m/s in the 10MWT for individuals with PD. With a 5% significance level and 80% power, 18 participants were required. Considering a 30% dropout rate, the final sample size was set at 26 (13 per group). However, this study will utilize an adaptive design and the sample size will be re-estimated using the effect sizes from the current study and recruitment will be adjusted accordingly. Between-group differences will be measured using a two-way repeated measures ANOVA, considering baseline, post-intervention, and follow-up assessments, following both intention-to-treat and per-protocol approaches (α=0.05).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of idiopathic PD confirmed by a neurologist
* classification between stages II to IV of the modified Hoehn & Yahr Scale (HY)
* use of anti-parkinsonian medication with stable pharmacological therapy for at least 6 months
* ability to walk independently in a 14-meter corridor with a walking speed ≤ 1.1 m/s
* ability to use a single-point cane during walking correctly and safely, and not being regular users of any type of assistive device since the diagnosis of PD.

Exclusion Criteria:

* cognitive impairment, assessed by the Mini Mental State Examination
* use deep brain stimulation,
* had any other neurological, cardiopulmonary or musculoskeletal condition that may compromise the tests performance

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in gait speed | At basilene (week 0), post-intervention (after the 3-week intervention), and one month after the cessation of the intervention (8-week follow-up).
  Gait speed will be measured by the 10-Meter Walk Test following previously described protocols

SECONDARY OUTCOMES:
Change from baseline in gait confidence | At basilene (week 0), post-intervention (after the 3-week intervention), and one month after the cessation of the intervention (8-week follow-up).
  Gait confidence will be assessed using the Gait Efficacy Scale-Brazil (mGES-Brazil). The mGES-Brazil is a ten-item scale that assesses an individual's confidence while walking in challenging circumstances.
Change from baseline in step length and cadence | At basilene (week 0), post-intervention (after the 3-week intervention), and one month after the cessation of the intervention (8-week follow-up).
  Step length and cadence will be assessed during the 10MWT following previously described protocols
Change from baseline in functional mobility | At basilene (week 0), post-intervention (after the 3-week intervention), and one month after the cessation of the intervention (8-week follow-up).
  Functional mobility will be assessed using the Timed "Up Go" test (TUG) following previously described protocols
Change from baseline in freezing of Gait | At basilene (week 0), post-intervention (after the 3-week intervention), and one month after the cessation of the intervention (8-week follow-up).
  Freezing of gait will be assessed by the Freezing of Gait Questionnaire (FOG-Q). This questionnaire has six items aimed at evaluating freezing during the gait in participants with PD. In addition to the questionnaire, the number and duration of freezing episodes that participants experience during the 10MWT and the TUG will be reported. The 10MWT and the TUG tests will be video recorded to allow detailed analysis of freezing episodes during the assessment.
Change from baseline in fear of falls | At basilene (week 0), post-intervention (after the 3-week intervention), and one month after the cessation of the intervention (8-week follow-up).
  Fear of falls will be assessed by the Falls Efficacy Scale - International (FES-I). This questionnaire has 16 items that assess the individual's concerns about the possibility of falling while carrying out different daily tasks
Satisfaction with using the cane | One month after the cessation of the intervention (8-week follow-up)
  Satisfaction regarding the use of the cane will be assessed by the Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0). The questionnaire has 12 items, scored from zero to five, where higher scores reflect greater participant satisfaction with assistive technology.

CONTACTS AND LOCATIONS:
Overall Officials: Christina DCM Faria, Doctor, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Federal University of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehdizadeh M, Martinez-Martin P, Habibi SA, Fereshtehnejad SM, Abasi A, Niazi Khatoon J, Saneii SH, Taghizadeh G. Reliability and Validity of Fall Efficacy Scale-International in People with Parkinson's Disease during On- and Off-Drug Phases. Parkinsons Dis. 2019 Jan 2;2019:6505232. doi: 10.1155/2019/6505232. eCollection 2019. PMID 30719277
- [Background] Keus S, Munneke M, Graziano M, et al. European Physiotherapy Guideline for Parkinson's disease. 2014; KNGF/ParkinsonNet, the Netherlands.
- [Background] Avelino, P. R., Menezes, K. K. P. de, Nascimento, L. R., Faria-Fortini, I., Faria, C. D. C. de M., Scianni, A. A., & Teixeira-Salmela, L. F. (2018). Adaptação transcultural da Modified Gait Efficacy Scale para indivíduos pós-acidente vascular encefálico. Revista de Terapia Ocupacional Da Universidade de São Paulo, 29(3), 230-236. https://doi.org/10.11606/issn.2238-6149.v29i3p230-236
- [Background] Mirelman A, Bonato P, Camicioli R, Ellis TD, Giladi N, Hamilton JL, Hass CJ, Hausdorff JM, Pelosin E, Almeida QJ. Gait impairments in Parkinson's disease. Lancet Neurol. 2019 Jul;18(7):697-708. doi: 10.1016/S1474-4422(19)30044-4. Epub 2019 Apr 8. PMID 30975519
- [Background] Kader M, Jonasson SB, Iwarsson S, Odin P, Nilsson MH. Mobility device use in people with Parkinson's disease: A 3-year follow-up study. Acta Neurol Scand. 2018 Jul;138(1):70-77. doi: 10.1111/ane.12942. Epub 2018 Apr 16. PMID 29658981
- [Background] Ni M, Hazzard JB, Signorile JF, Luca C. Exercise Guidelines for Gait Function in Parkinson's Disease: A Systematic Review and Meta-analysis. Neurorehabil Neural Repair. 2018 Oct;32(10):872-886. doi: 10.1177/1545968318801558. Epub 2018 Sep 28. PMID 30265211
- [Background] Bloem BR, Okun MS, Klein C. Parkinson's disease. Lancet. 2021 Jun 12;397(10291):2284-2303. doi: 10.1016/S0140-6736(21)00218-X. Epub 2021 Apr 10. PMID 33848468